CLINICAL TRIAL: NCT06400966
Title: The Effect of Jigsaw Technique on Childhood Epileptic Seizure Management Knowledge and Attitudes of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ayşe Kahraman, Assoc. Prof, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1919B012202144
Record Dates: First submitted 2024-04-27; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Jigsaw Technique; Epilepsy in Children; Nursing Student

STUDY DESIGN:
Intervention Model Description: The population of the research consisted of 173 3rd grade students who participated in the Child Health and Disease Nursing practice in the 2022-2023 academic year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Students in the Jigsaw technique group are divided into 5 home groups consisting of 8 people.Each student in the groups was randomly included to be an expert on a subject under 8 headings.In the home group, students assigned to different subject specializations were combined with students selected as experts in the same subject. This group was called the "expert group".The experts came together a week later, explained what they had learned on the common topic, discussed the topics they had taken notes while researching and reading in expert groups, and noted any additional points or missing parts they had learned. After completing their tasks in the expert groups, students returned to their home groups. They explained the information they learned in the expert group to each other in the home group, and as a home group, they brought together different topics and reported the main topic.
  Interventions: Other: Training method
- Traditional education group (No Intervention): Students in the traditional education group were given training by the researchers with a powerpoint presentation. Students are divided into 5 groups of 8 people. Training was given in 3 sessions for each group, for a total of 15 sessions. The training duration was 45 minutes for each session (one lesson hour).During the training, a projector, training slides and training videos on seizure types were used. Direct explanation and question-answer techniques were used in the training.

INTERVENTIONS:
Other: Training method — Jigsaw Technique
  Other Names: Jigsaw Technique
  Arms: Experimental

SUMMARY:
The aim of this study is to examine the effect of the education given to nursing students with the Jigsaw technique and traditional method on their knowledge and attitudes about childhood epileptic seizure management.

DETAILED DESCRIPTION:
It is important for nursing students, future health professionals, to gain sufficient professional knowledge and positive attitudes about epileptic seizure management in order to improve the quality of care they provide to children with epilepsy. Studies emphasize that the nursing education curriculum should focus more on education regarding epilepsy and epileptic seizures, and that different educational methods should be used to positively develop nursing students' knowledge and attitudes towards patients with epilepsy. One of the collaborative learning methods used in nursing education is the Jigsaw technique. Jigsaw technique is a student-centered and collaborative learning method that improves knowledge, skills and attitudes in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study

Exclusion Criteria:

* Not attending trainings and not filling out data collection forms

Ages: 20 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Childhood epilepsies and epileptic seizure management knowledge test scores | Before and after training (Half an hour before training and within half an hour after training)
  It consists of 15 questions answered as Yes-No-I Don't Know. The count was analyzed as a percentage. There is no total score.
Epilepsy knowledge and attitude scale scores | Before and after training (Half an hour before training and within half an hour after training)
  Epilepsy Knowledge and Attitude Scale consists of 16 items measuring knowledge about epilepsy and 14 items measuring attitude. For the knowledge scale, correct = 1, incorrect and no idea = 0. A high score indicates high knowledge. Responses regarding the attitude part of the scale; I strongly disagree = 5, I disagree = 4, I have no idea = 3, I agree = 2, and I completely agree = 1. Higher scores indicate a more positive attitude towards epilepsy.

SECONDARY OUTCOMES:
Students' self-confidence | Before and after training (Half an hour before training and within half an hour after training)
  Students were determined based on self-report. It was answered as Yes or No.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Nursing, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No